CLINICAL TRIAL: NCT03090035
Title: Impact of Interleukin 28B (rs12979860) Genotype on Virological Responses in Chronic Hepatitis C Treatment
Brief Title: Impact of Interleukin 28B (rs12979860) Genotype on Virological Responses Chronic Hepatitis C Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sheikh Zayed Medical College (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: sheikhZMC
Record Dates: First submitted 2017-02-27; First posted 2017-03-24 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Hepatitis C; Hepatitis C Relapse
Keywords: HCV genotype 2, HCV genotype 3, IL-28B, PEG-INF.
MeSH Terms: conditions — Hepatitis C | interventions — Ribavirin

STUDY DESIGN:
Intervention Model Description: Clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- chronic hepatitis C genotype 2 or 3 (Experimental): In all patients Pegylated Interferon α2 (pegIFN) plus Ribavirin were given in standard doses. Peg-INF was given in a dose of 180 μg/week and ribavirin 1200 mg/day to every patient for the period of 24 weeks for HCV genotype 2 & 3
  Interventions: Drug: Pegylated Interferon α2; Drug: Ribavirin

INTERVENTIONS:
Drug: Pegylated Interferon α2 — Peg-INF was given in a dose of 180 μg/week
  Other Names: Unipg
Drug: Ribavirin — ribavirin 1200 mg/day to every patient for the period of 24 weeks for HCV genotype 2 & 3
  Other Names: Ribavil

SUMMARY:
Objective:

Pegulated Interferon α2 plus ribavirin is a treatment of choice in patients with chronic hepatitis C infection. This study was conducted to find out the frequency of different IL-28B (rs12979860) genotypes in patients with chronic hepatitis C (HCV genotype type 2 & 3) infection treated with Pegulated Interferon α2 plus ribavirin and to evaluate the role of IL-28B genotypes in achieving Sustained Virological Response (SVR).

Methods:

In this non-randomized observational study, ninety eight (98) patients with diagnosis of chronic hepatitis C were included. In all patients, Peg-IFN plus Ribavirin were given in standard doses for 24 weeks. End treatment response, sustained virological response, and relapse rate were the primary endpoints of this study. Analysis of IL28B (rs12979860) polymorphism (CC, CT and TT) was performed by PCR-RFLP protocol.

DETAILED DESCRIPTION:
INTRODUCTION:

Hepatitis C virus (HCV) is a major health problem that effects nearly 170 million people worldwide [1, 2]. According to a report, about 64-103 million people are suffering from chronic HCV infection [3] and this chronic infection results in liver scarring, hepatocellular carcinoma or end-stage liver disease in about forty thousand (40,000) patients every year [4, 5]. According to WHO, liver disease initiated by chronic hepatitis C infection is responsible for more than 35 thousand deaths and 3 to 4 million people are infected every year[3, 6]. Hepatitis C Virus has been classified into seven genotypes and several subtypes, which are associated with distinct forms of geographic dispersal [7, 8]. The success of HCV treatment is affected by many viral, treatment or host factors.

Pegulated Interferon α2 plus ribavirin is a treatment of choice in patients with chronic hepatitis C infection. Sustained virological response (SVR) rate with this treatment in HCV-2 & 3 has been reported to be 58-84% in previously untreated patients [9]. SVR can be affected by liver cirrhosis, hepatocellular carcinoma, ethnicity, age, gender and obesity. [10, 11] It has been clarified by some studies that interleukin-28B has an important role in the treatment success of HCV infection and IL-28B CC genotype is associated with 2 folds higher sustained virological response (SVR) as compared to CT and TT genotype [12-14]. The aim of present study was to find out the frequency of different IL28B (rs12979860) genotypes in patients with chronic hepatitis C (genotype type 2 or 3) infection treated with Pegulated Interferon α2 plus ribavirin and to evaluate the role of IL-28B genotypes in achieving Sustained Virological Response (SVR).

METHODS:

This non-randomized observational study was conducted in Sheikh Zayed Medical College/Hospital Rahim Yaar Khan. A total of ninety eight (98) patients with diagnosis of chronic hepatitis C genotype 2 or 3 were involved in this study. The duration of study was from January 2015 to January 2016. People living in Rahim Yaar Khan City belongs to different ethinic backgrounds because this city is located at the junction of three provinces of Pakistan (total provinces are four), so people residing here represent the whole Pakistani population living in different provinces. Institutional ethical approval was taken before starting this research work. A written informed consent was taken from every patient before including him/her in this study.

The diagnosis of chronic hepatitis C was made through liver enzyme levels, HCV-RNA positivity and anti-HCV antibody test. Patients with other chronic liver disorders, with positive hepatitis B virus (HBV), and human immunodeficiency virus (HIV) infection were excluded from this study.

Treatment Protocol and Detection of IL28B Polymorphism:

In all patients Pegulated Interferon α2 (pegIFN) plus Ribavirin were given in standard doses. PegINF was given in a dose of 180 μg/week and ribavirin 1200 mg/day to every patient for the period of 24 weeks for HCV genotype 2 & 3.

PCR analysis was done in every patient before starting the treatment, after 24 weeks of treatment (to see end treatment response) and 48 weeks (to evaluate SVR and relapse rate) of treatment. Analysis of IL28B (rs12979860) polymorphism (CC, CT and TT) was performed by PCR restriction fragment length polymorphism (RFLP) assay protocol. Pyrosequencing method was used to determine HCV genotypes.

Data analysis was done using SPSS V17 software. Mean and standard deviation were used for the presentation of quantitative variables. Frequency and percentages were used to present qualitative data. Chi-square test/Fisher Exact test was used to compare qualitative data. P-value <0.05 was taken as significant.

ELIGIBILITY:
Inclusion Criteria:

* patients with diagnosis of chronic hepatitis C genotype 2 or 3

Exclusion Criteria:

* Patients with hepatitis genotype I and IV

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2014-07-01 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
Treatment Success rate | after 24 weeks of treatment
  Treatment Success rate (End Treatment Response) was noted to check the adequency of treatment

SECONDARY OUTCOMES:
Sustained Virological Response | After 48 weeks of treament
  Sustained Virological Response was noted to check treatment success after extended period
Relapse Rate | After 48 weeks of treament
  Relapse Rate to check re-occurrence of Hepatitis infection

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad ZM Babar, FCPS, Principal Investigator — Sheikh Zayed Medical College/Hospital
Locations (1):
- Muhammad Zafar Majeed Babar, Sadiqabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shepard CW, Finelli L, Alter MJ. Global epidemiology of hepatitis C virus infection. Lancet Infect Dis. 2005 Sep;5(9):558-67. doi: 10.1016/S1473-3099(05)70216-4. PMID 16122679
- [Result] Wantuck JM, Ahmed A, Nguyen MH. Review article: the epidemiology and therapy of chronic hepatitis C genotypes 4, 5 and 6. Aliment Pharmacol Ther. 2014 Jan;39(2):137-47. doi: 10.1111/apt.12551. Epub 2013 Nov 19. PMID 24251930
- [Result] Gower E, Estes C, Blach S, Razavi-Shearer K, Razavi H. Global epidemiology and genotype distribution of the hepatitis C virus infection. J Hepatol. 2014 Nov;61(1 Suppl):S45-57. doi: 10.1016/j.jhep.2014.07.027. Epub 2014 Jul 30. PMID 25086286
- [Result] Wise M, Bialek S, Finelli L, Bell BP, Sorvillo F. Changing trends in hepatitis C-related mortality in the United States, 1995-2004. Hepatology. 2008 Apr;47(4):1128-35. doi: 10.1002/hep.22165. PMID 18318441
- [Result] Ghany MG, Strader DB, Thomas DL, Seeff LB; American Association for the Study of Liver Diseases. Diagnosis, management, and treatment of hepatitis C: an update. Hepatology. 2009 Apr;49(4):1335-74. doi: 10.1002/hep.22759. No abstract available. PMID 19330875
- [Result] Chen SL, Morgan TR. The natural history of hepatitis C virus (HCV) infection. Int J Med Sci. 2006;3(2):47-52. doi: 10.7150/ijms.3.47. Epub 2006 Apr 1. PMID 16614742
- [Result] Argentini C, Genovese D, Dettori S, Rapicetta M. HCV genetic variability: from quasispecies evolution to genotype classification. Future Microbiol. 2009 Apr;4(3):359-73. doi: 10.2217/fmb.09.8. PMID 19327119
- [Result] Smith DB, Bukh J, Kuiken C, Muerhoff AS, Rice CM, Stapleton JT, Simmonds P. Expanded classification of hepatitis C virus into 7 genotypes and 67 subtypes: updated criteria and genotype assignment web resource. Hepatology. 2014 Jan;59(1):318-27. doi: 10.1002/hep.26744. PMID 24115039
- [Result] Yee BE, Nguyen NH, Zhang B, Lin D, Vutien P, Wong CR, Lutchman GA, Nguyen MH. Sustained virological response and its treatment predictors in hepatitis C virus genotype 4 compared to genotypes 1, 2, and 3: a meta-analysis. BMJ Open Gastroenterol. 2015 Jul 9;2(1):e000049. doi: 10.1136/bmjgast-2015-000049. eCollection 2015. PMID 26462288
- [Result] Chen TY, Hsieh YS, Wu TT, Yang SF, Wu CJ, Tsay GJ, Chiou HL. Impact of serum levels and gene polymorphism of cytokines on chronic hepatitis C infection. Transl Res. 2007 Aug;150(2):116-21. doi: 10.1016/j.trsl.2007.01.007. Epub 2007 May 23. PMID 17656331
- [Result] Younossi ZM, McCullough AJ. Metabolic syndrome, non-alcoholic fatty liver disease and hepatitis C virus: impact on disease progression and treatment response. Liver Int. 2009 Mar;29 Suppl 2:3-12. doi: 10.1111/j.1478-3231.2008.01949.x. PMID 19187068
- [Result] Ge D, Fellay J, Thompson AJ, Simon JS, Shianna KV, Urban TJ, Heinzen EL, Qiu P, Bertelsen AH, Muir AJ, Sulkowski M, McHutchison JG, Goldstein DB. Genetic variation in IL28B predicts hepatitis C treatment-induced viral clearance. Nature. 2009 Sep 17;461(7262):399-401. doi: 10.1038/nature08309. Epub 2009 Aug 16. PMID 19684573
- [Result] Grebely J, Petoumenos K, Hellard M, Matthews GV, Suppiah V, Applegate T, Yeung B, Marks P, Rawlinson W, Lloyd AR, Booth D, Kaldor JM, George J, Dore GJ; ATAHC Study Group. Potential role for interleukin-28B genotype in treatment decision-making in recent hepatitis C virus infection. Hepatology. 2010 Oct;52(4):1216-24. doi: 10.1002/hep.23850. PMID 20803561
- [Result] Tanaka Y, Nishida N, Sugiyama M, Kurosaki M, Matsuura K, Sakamoto N, Nakagawa M, Korenaga M, Hino K, Hige S, Ito Y, Mita E, Tanaka E, Mochida S, Murawaki Y, Honda M, Sakai A, Hiasa Y, Nishiguchi S, Koike A, Sakaida I, Imamura M, Ito K, Yano K, Masaki N, Sugauchi F, Izumi N, Tokunaga K, Mizokami M. Genome-wide association of IL28B with response to pegylated interferon-alpha and ribavirin therapy for chronic hepatitis C. Nat Genet. 2009 Oct;41(10):1105-9. doi: 10.1038/ng.449. Epub 2009 Sep 13. PMID 19749757